CLINICAL TRIAL: NCT00906646
Title: Preparation of Patients for Cardiac Surgery
Acronym: MPM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Griffith University (Other)
Responsible Party: Professor Franklin Rosenfeldt, Alfred Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91/04
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Artery Bypass Graft Surgery; Cardiac Valve Surgery
Keywords: cardiac; surgery; metabolic; supplements; antioxidant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metabolic therapy (Experimental): Metabolic therapy with antioxidants and cellular energisers
  Interventions: Dietary Supplement: Metabolic therapy
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Metabolic therapy — Coenzyme Q10 - 100 mg tds Magnesium orotate - 400 mg tds Lipoic acid - 100 mg tds Omega-3 fatty acids - 300 mg (in 1 g fish oils) tds Selenium - 200 µg
  Arms: Metabolic therapy
Dietary Supplement: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This was a prospective randomised trial of metabolic therapy including antioxidants and cellular energisers to determine whether this therapy could improve the results of cardiac surgery. The hypothesis was that the metabolic therapy could improve clinical recovery.

DETAILED DESCRIPTION:
Objective Perioperative therapy with antioxidants and metabolic substrates has the potential to reduce oxidative stress and improve recovery from cardiac surgery, particularly in elderly and high risk cases. The aim of the study was to assess the effect of perioperative metabolic therapy at a biochemical and clinical level in cardiac surgical patients.

Methods Patients (n = 117, mean age 65 ± 1.0 years, 74% male) undergoing elective coronary artery bypass graft (CABG) and/or valve surgery were randomized to receive for a minimum of 2 weeks before and one month after surgery, either metabolic therapy (coenzyme Q10, magnesium orotate, lipoic acid, omega-3 fatty acids and selenium) or placebo. Biochemical and clinical outcomes were assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective coronary artery bypass graft (CABG) and/or valve surgery

Exclusion Criteria:

* urgent or emergency surgery
* NYHA class IV heart failure
* taken antioxidant supplements in the previous month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2004-04; Primary Completion 2006-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Troponin release | 24 hours after surgery

SECONDARY OUTCOMES:
Length of hospital stay | 1 month
Rate of atrial fibrillation | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franklin L Rosenfeldt, MBBS, MD, Study Director — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia